CLINICAL TRIAL: NCT02589093
Title: Validation of a Nociception Monitor in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Philippe Richebé, M.D., Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14074
Record Dates: First submitted 2015-10-25; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: Analgesia; Monitoring; Analgesia Nociception Index; ANI; PhysioDoloris; Pain
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stimulation (Experimental): Subjects will receive progressive electrical stimulations with an external nerve stimulator over the ulnar nerve, from 0 mA to 30 mA in increments of 5 (2 Hz single twitch mode), for 3 minutes at each intensity. They will be asked to score their pain level (NRS 0-10) every minute. ANI will be recorded constantly.
  Interventions: Device: Stimulation

INTERVENTIONS:
Device: Stimulation

SUMMARY:
Anesthesiology daily practice consists in management of sedation, immobility and analgesia. The monitoring of this last component remains largely based on indirect signs with poor sensitivity and specificity such as heart rate and blood pressure. Accordingly, there is an increased demand for more accurate analgesia monitors. Several parameters have been studied in the recent years such as spectral entropy, skin conductance, pupillometry or heart rate variability (HRV). The HRV is influenced by the balance of sympathetic and parasympathetic tones, and is therefore influenced by pain and analgesia.

MDoloris Medical Systems SAS, located in Lille, France, had developed a monitor called PhysioDoloris (TM) that uses an analysis of the HRV to generate a clinically useable index, the Analgesia-Nociception Index (ANI). The ANI varies from 0 to 100, a lower number indicating less parasympathetic tone. It has been shown in previous studies under general anesthesia to decrease at the moment of surgical incision and pneumoperitoneum inflation and to increase with opioids administration.

The purpose of this study is to show a correlation between the variation of the ANI with pain scores in awake healthy volunteers who are subjected to standardized painful stimuli of increasing intensity. The investigators hypothesize that an increasing pain score will correlate with decreasing ANI values.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18-80 years old

Exclusion Criteria:

* Heart disease
* Neurological disease
* Allergy to cutaneous electrodes
* Chronic pain and/or chronic analgesics consumption
* Medication affecting the autonomic nervous system
* Inability to understand a numeric rating scale (NRS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
ANI index values during increasing intensities of moderately painful electrical stimulation at the forearm level. | Assessed during the entire cycle of stimulation (approx. 30 min)
  The ANI is an index that can vary from 0 (maximum pain) to 100 (no pain) in humans. The primary objective of this study will be to record the ANI values all along the time period of the clinical evaluation, while the subjects are submitted to standardized electrical stimulation going from 0 mA (no stimulation) to a maximum of 25 mA (or less according to the subject tolerance).
  Each stimulation lasts for 3 minutes. During these 3 minutes the ANI is electronically recorded automatically but the Physiodoloris device. The quantitavive value of the index is then analyzed during each stimulation and for all the stimulations.
  This will allow to evaluate whether it exists any correlation between the ANI values and the intensity of the electrical stimulation.

SECONDARY OUTCOMES:
ANI correlation with Numerical Rating Scale (NRS) of pain | Assessed during the entire cycle of stimulation (approx. 30 min)
  NRS and ANI absolute values will be recorded all along the study duration (approx. 30min). This will allow to evaluate a likely correlation between the ANI absolute values and the NRS values.
Heart rate correlation with ANI | Assessed during the entire cycle of stimulation (approx. 30 min)
  ANI values and HR are recorded for the whole duration of the study. A correlation between these two criteria will be evaluated to know if HR increases (more pain) when ANI decreases (more pain).
Blood pressure correlation with ANI | Assessed during the entire cycle of stimulation (approx. 30 min)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebé, M.D., Principal Investigator — Maisonneuve-Rosemont Hospital

REFERENCES:
- [Derived] Issa R, Julien M, Decary E, Verdonck O, Fortier LP, Drolet P, Richebe P. Evaluation of the analgesia nociception index (ANI) in healthy awake volunteers. Can J Anaesth. 2017 Aug;64(8):828-835. doi: 10.1007/s12630-017-0887-z. Epub 2017 Apr 21. PMID 28432612